CLINICAL TRIAL: NCT02578069
Title: A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Efficacy of the NOVA Sirolimus Eluting Stent Versus the Apollo Stent
Brief Title: First-in-man Trial Evaluating the Safety and Efficacy of the NOVA Intracranial Stent (NOVA Trial)
Acronym: NOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOVA-001
Record Dates: First submitted 2015-09-29; First posted 2015-10-16 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2019-01

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Intracranial Stenting
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): NOVA Intracranial sirolimus eluting stent system
  Interventions: Device: NOVA Intracranial Sirolimus Eluting Stent System
- Control (Active Comparator): Apollo Intracranial stent system
  Interventions: Device: Apollo Intracranial Stent System

INTERVENTIONS:
Device: NOVA Intracranial Sirolimus Eluting Stent System — A sirolimus eluting intracranial stent system with polylactic-co-glycolic acid (PLGA) biodegradable drug carrier and electro-grated polybutyl methacrylate (PBMA) base coating. The stent platform is made of 316L stainless steel.
  Arms: Experimental
Device: Apollo Intracranial Stent System — A 316L stainless steel balloon-expandable intracranial stent system
  Arms: Control

SUMMARY:
Prospective, multi-center, randomized 1:1 single blind trial using NOVA sirolimus eluting stent versus Apollo bare metal stent conducted in approximately 15 interventional neurology centers in China. The study was sponsored by Sino Medical Sciences Technology Inc.

DETAILED DESCRIPTION:
The study will enroll 264 subjects overall in two groups (randomized 1:1). The study follow-up will occur at 1, 6 and 12 months post-stent implantation. All patients will undergo angiography assessment (DSA/CTA) at 12 months follow-up. Angiography assessment will be performed at baseline (pre- and post-procedure) and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age;
2. Primary or recurrent symptomatic intracranial arteriostenosis through the internal medicine treatment (i.e. stroke or transient ischemic attack within 90 days during the treatment with at least one anti-thrombotic drugs and vascular risk factor intervention e.g. hypertensors for hypertension and hypolipidemics for hyperlipidemia);
3. No transient ischemic attack (TIA) or ischemic stroke occurred within 2 weeks prior to stenting procedure;
4. ≥70% stenosis of intracranial responsible vessel under the DSA angiography (as judged through the WASID method);
5. Poor blood circulation in the side branch of responsible vessel area under the angiography within one week prior to stenting procedure:

   Score of blood circulation in the side branch under the DSA <3 or blood flow rate peak ≥200cm/s at the systolic phase under the transcranial doppler ultrasonic examination (TCD); or no apparent side branch compensation in the responsible vessel area under CTA or score of blood circulation in the side branch under the CTA <2;
6. The target lesion reference diameter must be visually estimated to be ≥2.0 mm in diameter, and lesion length must be <15 mm; no lesion observed in the distal vessel;
7. Atherosclerosis lesions;
8. mRS < 3;
9. Written informed consent.

Exclusion Criteria:

1. >70% intracranial large-vessel stenosis beyond the responsible vessel;
2. >70% stenosis observed at the intracranial large-vessel distal to the responsible vessel or >70% stenosis observed at the intracranial/extracranial large-vessel proximal to the responsible vessel;
3. Acute ischemic stroke within 3 weeks;
4. Obstruction of perforating branch artery under the skull MRI;
5. Intracranial hemorrhage in the angiopathic area within 6 weeks;
6. Patient was treated by thrombolytic therapy within 24 hours;
7. Patients underwent surgery within 30 days or plan for surgery within 3 months post-stenting procedure;
8. Severe calcified lesions;
9. Patients have been treated by intracranial/extracranial stenting procedures prior to this study;
10. Nonatherosclerosis lesions;
11. Patients with potential sources for cardiac embolism;
12. Concomitant intracranial tumor, aneurysm or intracranial arteriovenous malformation;
13. Known hypersensitivity or contraindication to aspirin, heparin, antiplatelet medication specified for use in the study, sirolimus, poly(lactic-co-glycolic acid) polymers, or poly(n-butyl methacrylate);
14. Hemoglobin <100g/L, platelet count <100,000 cells/mm3, International normalized ratio (INR) >1.5 (irreversible) or uncorrectable hemorrhagic factors;
15. Serious neural dysfunction due to the responsible angiopathy as the sequel of cerebral infarction (mRS≥3);
16. Known liver or renal insufficiency (ALT> 3x upper limit or AST > 3x upper limit, creatinine > 1.5x upper limit);
17. Life expectancy < 2 years;
18. Pregnant/lactating female patients;
19. Patients with cognitive impairment or mental diseases;
20. The patient participated in another investigational device or drug study within 3 months;
21. Inapplicable for intravascular stenting treatment as per investigators judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
In stent restenosis rate (> 50% restenosis) | 12 months post-procedure
  Angiography assessment at 12 months post-procedure

SECONDARY OUTCOMES:
Stroke and death events | within 30 days after stenting
Target vessel ischemic stroke event | between 30 days and 1 year post-procedure
Acute procedural success rate (stenosis < 30%) | 1 year
Target vessel stroke or death events | within 30 days after stenting
Non-target vessels ischemic stroke event | between 30 days and 1 year post-procedure
Recurrent ischemic stroke in the involved vascular area | between 30 days and 1 year post-procedure
Cerebral parenchyma hemorrhage, subarachnoid hemorrhage and intraventricular bleeding events | between 30 days and 1 year post-procedure
Death event | between 30 days and 1 year post-procedure
Transient ischemic attack event | within 1 year post-procedure
National Institutes of Health Stroke Scale (NIHSS) evaluation | at 1 and 12 months
modulate RANK score （mRS）evaluation | at 1 and 12 months
Montreal Cognitive Assessment (MoCA) evaluation | at 1 and 12 months
EQ-5D score evaluation | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

REFERENCES:
- [Derived] Jia B, Zhang X, Ma N, Mo D, Gao F, Sun X, Song L, Liu L, Deng Y, Xu X, Zhang Y, Liu Z, Guan S, Zhang F, Li B, Zheng H, Liu X, Liu Y, Chen K, Shuai J, Wan J, Wang J, Shi X, Li T, Chang B, Liebeskind DS, Yu W, Miao Z; NOVA Trial Investigators. Comparison of Drug-Eluting Stent With Bare-Metal Stent in Patients With Symptomatic High-grade Intracranial Atherosclerotic Stenosis: A Randomized Clinical Trial. JAMA Neurol. 2022 Feb 1;79(2):176-184. doi: 10.1001/jamaneurol.2021.4804. PMID 34982098